CLINICAL TRIAL: NCT02016677
Title: An Observational Study Exploring the Esthetic Outcomes of Breast Reduction Surgery and /or Mastopexy
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment rate. Low scientific value
Sponsor: Orbix Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLI-02
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-10

CONDITIONS: Macromastia
Keywords: Breast reduction; Mastopexy; Sagging
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- observation: no specific treatment. Long term observation the results of any breast lifting or reduction surgeries

SUMMARY:
The purpose of the study is to collect data regarding the aesthetic outcomes of patients who had breast reduction surgery and /or mastopexy in terms such as scaring, patient satisfaction, breast ptosis assessment including taking photographs and filling questionnaires.

DETAILED DESCRIPTION:
This is a prospective observational study, single center cohort to explore the aesthetic outcomes of patients who had breast reduction and / or mastopxy surgery. The surgical intervention will be determined by the clinician with no correlation to this study.

The study will focus on the aesthetic aspects of the clinical outcome resultant from the breast surgery in par course of 5 years. Scar tissue assessment and patient's reported data (satisfaction and well-being) will be collected.

Suitable patients will be assessed for study eligibility at a screening visit and, if eligible, will be scheduled for breast surgery according to the patient and surgeon discretion.

At each follow up visit, patients will undergo clinical general examination, breast and ptosis endearments, scar appearance , aesthetic evaluation. Patients will fill satisfaction questionnaires

ELIGIBILITY:
Inclusion Criteria:

1. Female patient older than 30 years of age.
2. Patients willing to participate as evidenced by signing the written informed consent.
3. Patient that was found by her physician illegible for breast reduction surgery and /or mastopxy

Exclusion Criteria:

1. Active psychiatric illness, cognitive or sensory impairment. 2. Physical impairment that may prevent filling out a paper and pencil survey or responding to interview questions

-

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female Patients, 30 years of age or older referred for elective breast reduction surgery and /or mastopxy
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Measuring the aesthetic outcomes of pre /post- surgical breast ptosis | during 5 years post- surgically
  Breast measurements consists on:
  * Breast cup size
  * Distortions or skin retractions
  * Symmetry between the two breasts
  * Ptosis grade evaluated on the basis of an I-IV scale
  * Methods to measure breast shape and symmetry
  * Skin texture (soft or hard)
  * Skin consistency
  * Nipple location on the breast mound scored on a scale of 1 - 5
  * Areola diameter (mm)
  * The shape of the breast scored on a scale of 1 - 5
  * Scar Appearance evaluation -VAS score
  * Patient satisfaction questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Arik Zaretski, MD, Study Director — TASMC
Locations (1):
- The Plastic Surgery Department The Tel Aviv Sourasky Medical Center, Tel Aviv, Israel